CLINICAL TRIAL: NCT02905175
Title: Porphyromonas Gingivalis Contribution in Rheumatoid Arthritis (RA).
Brief Title: Rheumatoid Arthritis Patients and Porphyromonas Gingivalis
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1408022; 2014-A01688-39 (Other: ANSM)
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Last update posted 2019-07-26 (Actual); Status verified 2018-10

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; Porphyromonas gingivalis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sample and synovial tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rheumatoid arthritis: blood sample specimen and synoviocytes from synovial tissue
  Interventions: Procedure: blood sample; Procedure: synovial tissue
- Osteoarthritis: blood sample specimen and synoviocytes from synovial tissue
  Interventions: Procedure: blood sample; Procedure: synovial tissue

INTERVENTIONS:
Procedure: blood sample
Procedure: synovial tissue — synoviocytes from synovial tissue

SUMMARY:
Rheumatoid arthritis (RA) is the most frequent joint inflammatory disease inducing joint destruction strongly correlated with anti-citrullinated protein antibodies citrullinated anti-peptide (ACPA). Precise RA etiology remained unclear with a described association between RA and periodontal disease. The missing link could be a gram-negative anaerobic bacterium called Porphyromonas gingivalis (P. gingivalis), which is heavily involved in periodontal disease and able to induce gingival citrullinated protein via an enzyme called peptidyl arginine deiminase (PAD). DNA of P. gingivalis was detected in synovial tissue and in peripheral blood mononuclear cell. To improve knowledge of P. gingivalis involvement in RA, the investigators will compare its effect on various cell type with comparison with another oral bacteria Provatella intermedia.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 ans
* RA or osteoarthritis with joint surgery planned
* Informed consent approved and signed

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatoid arthritis and osteoarthritis
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2016-01-13 (Actual); Primary Completion 2016-06-27 (Actual); Study Completion 2016-06-27 (Actual)

PRIMARY OUTCOMES:
Comparison of genetic signature after induction by P. gingivalis and P. intermedia on synoviocytes | day 1

SECONDARY OUTCOMES:
Comparison of specific transcriptome profile induced by P. gingivalis compared to P. intermedia on peripheral blood mononuclear cells (PBMC) and gingival fibroblasts | day 1
Comparison of transcriptome profile between P. gingivalis and P. intermedia on RA synovial cells. | day 1
Comparison of the transcriptomic profile between RA and osteoarthritis synoviocytes | day 1

CONTACTS AND LOCATIONS:
Overall Officials: Hubert Marotte, phD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No